CLINICAL TRIAL: NCT04164563
Title: A Randomized Controlled Trial of Non-Operative Ankle Fractures: Even-Up Orthotic Shoe Lift and CAM Walking Boot Wear
Brief Title: Even-Up to Minimize Secondary Site Pain For Ankle Fracture
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: We have elected to discontinue enrolling patients.
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Jeremy Smith, Assistant Professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2019P002694
Record Dates: First submitted 2019-11-13; First posted 2019-11-15 (Actual); Results first posted 2022-10-18 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-09

CONDITIONS: Arthralgia; Trouble Balancing
Keywords: Joint pain; Ankle fracture; Leg length discrepancy; CAM boot; Even-Up
MeSH Terms: conditions — Arthralgia; Ankle Fractures; Leg Length Inequality

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Masking Description: Both patients and providers are aware that patients are being assigned to either control or experimental group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Control (No Intervention): Standard CAM boot treatment without Even-Up device.
- Study (Experimental): CAM boot treatment with Even-Up for contralateral extremity.
  Interventions: Device: Even-Up

INTERVENTIONS:
Device: Even-Up — Orthotic shoe lift worn on contralateral foot to increase leg length
  Arms: Study

SUMMARY:
Evaluating impact of use of Even-Up shoe wear device for patients treated in CAM boot walker for an ankle fracture. Randomized controlled trial, randomizing patients into control group with boot treatment only versus boot treatment with Even-Up device on contralateral extremity.

DETAILED DESCRIPTION:
A variety of foot and ankle injuries can be treated effectively through the use of a controlled ankle movement (CAM) walker boot. CAM walker boots protect the injured area by restricting foot and ankle motion, providing a stable platform to distribute forces while bearing weight, and allowing the user to rollover the foot during ambulation because of a rocker bottom-shaped sole. Such qualities lend the CAM walker boot to provide ankle support that can be advantageous compared with other commonly used methods. Despite their utility, CAM walker boots create a simulated leg-length discrepancy (LLD), which can result in altered biomechanics during ambulation. Additionally, a LLD can be associated with lower back and joint pain.

We have previously conducted a study that suggests a relationship exists between CAM walker boot treatment and pain at sites other than the extremity being treated. There have been several randomized controlled trials (RCTs) examining a relationship between the correction of inherent LLD with insole inserts and lower back pain. Furthermore, there has been a past RCT and there is a current RCT examining a relationship between the use of the EVENup orthotic shoe lift to correct CAM walker boot simulated LLD and pain at sites other than the extremity being treated. However, these studies were not conducted with patient populations with uniform injuries. To the best of our knowledge, an RCT has not been conducted with the EVENup orthotic shoe lift to examine this relationship in a uniform patient population with nonoperative ankle fractures. This RCT aims to assess the efficacy of the EVENup orthotic shoe lift, towards reducing and even preventing such pain that may be associated with this common course of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Non-operative Treatment of Ankle Fracture
* CAM boot as treatment for injury
* Weight bearing ad lib

Exclusion Criteria:

* Pregnancy
* Non-English speaking
* Recent surgery for lower extremity or back
* Recent other injury to lower extremity or back
* Restricted weight bearing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-11-14 (Actual); Primary Completion 2020-09-10 (Actual); Study Completion 2020-09-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy T Smith, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Waverly BJ, Sorensen MD, Sorensen TK. Early Weightbearing Protocol in Operative Fixation of Acute Jones Fractures. J Foot Ankle Surg. 2018 May-Jun;57(3):489-493. doi: 10.1053/j.jfas.2017.11.005. PMID 29685559
- [Background] DiGiovanni BF, Moore AM, Zlotnicki JP, Pinney SJ. Preferred management of recalcitrant plantar fasciitis among orthopaedic foot and ankle surgeons. Foot Ankle Int. 2012 Jun;33(6):507-12. doi: 10.3113/FAI.2012.0507. PMID 22735325
- [Background] Mittal R, Harris IA, Adie S, Naylor JM; CROSSBAT Study Group. Surgery for Type B Ankle Fracture Treatment: a Combined Randomised and Observational Study (CROSSBAT). BMJ Open. 2017 Mar 27;7(3):e013298. doi: 10.1136/bmjopen-2016-013298. PMID 28348185
- [Background] Simpson MR, Howard TM. Tendinopathies of the foot and ankle. Am Fam Physician. 2009 Nov 15;80(10):1107-14. PMID 19904895
- [Background] Vulcano E, Deland JT, Ellis SJ. Approach and treatment of the adult acquired flatfoot deformity. Curr Rev Musculoskelet Med. 2013 Dec;6(4):294-303. doi: 10.1007/s12178-013-9173-z. PMID 23765382
- [Background] Ready LV, Fisk EG, Ciurylo W, Chiodo CP, Bluman EM, Smith JT. Associated Joint Pain With Controlled Ankle Movement Walker Boot Wear. J Am Acad Orthop Surg Glob Res Rev. 2018 Nov 27;2(12):e044. doi: 10.5435/JAAOSGlobal-D-18-00044. eCollection 2018 Dec. PMID 30680366
- [Background] Keene DJ, Willett K, Lamb SE. The Immediate Effects of Different Types of Ankle Support Introduced 6 Weeks After Surgical Internal Fixation for Ankle Fracture on Gait and Pain: A Randomized Crossover Trial. J Orthop Sports Phys Ther. 2016 Mar;46(3):157-67. doi: 10.2519/jospt.2016.6212. Epub 2016 Jan 26. PMID 26813753
- [Background] White SC, Gilchrist LA, Wilk BE. Asymmetric limb loading with true or simulated leg-length differences. Clin Orthop Relat Res. 2004 Apr;(421):287-92. doi: 10.1097/01.blo.0000119460.33630.6d. PMID 15123962
- [Background] O'Toole GC, Makwana NK, Lunn J, Harty J, Stephens MM. The effect of leg length discrepancy on foot loading patterns and contact times. Foot Ankle Int. 2003 Mar;24(3):256-9. doi: 10.1177/107110070302400310. PMID 12793490
- [Background] Subotnick SI. Limb length discrepancies of the lower extremity (the short leg syndrome). J Orthop Sports Phys Ther. 1981;3(1):11-6. doi: 10.2519/jospt.1981.3.1.11. PMID 18810144
- [Background] Rannisto S, Okuloff A, Uitti J, Paananen M, Rannisto PH, Malmivaara A, Karppinen J. Correction of leg-length discrepancy among meat cutters with low back pain: a randomized controlled trial. BMC Musculoskelet Disord. 2019 Mar 14;20(1):105. doi: 10.1186/s12891-019-2478-3. PMID 30871549
- [Background] Defrin R, Ben Benyamin S, Aldubi RD, Pick CG. Conservative correction of leg-length discrepancies of 10mm or less for the relief of chronic low back pain. Arch Phys Med Rehabil. 2005 Nov;86(11):2075-80. doi: 10.1016/j.apmr.2005.06.012. PMID 16271551
- [Background] Kipp D, Village D, Edwards KJ. Effectiveness of Evenup Shoe-Lift Use Among Individuals Prescribed a Walking Boot. J Allied Health. 2017 Summer;46(2):104-110. PMID 28561867
- See also: Study of an Orthotic Designed to Equalize Leg Lengths for Patients with Injuries Managed in Walking Boots — http://clinicaltrials.gov/ct2/show/NCT03848949

RESULTS

PARTICIPANT FLOW:
Groups:
- Group I: CAM Walker Boot: Patients in Group I were assigned to receive a course of CAM walker boot treatment for a period of six weeks.
- Group II: CAM+EVENup Orthotic Shoe Lift: Patients in Group II were assigned to receive a course of CAM walker boot treatment with an EVENup orthotic shoe lift to be worn on the contralateral foot for a period of six weeks.
Period: Overall Study
Arm/Group | Group I: CAM Walker Boot | Group II: CAM+EVENup Orthotic Shoe Lift
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group I: CAM Walker Boot | Group II: CAM+EVENup Orthotic Shoe Lift | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 6
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36 (17.1) | 48 (21.9) | 42 (18.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 3 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 6
FAAM (0 - 100) [Mean (Standard Deviation); unit: units on a scale] — FAAM-ADL (Foot and Ankle Ability Measure - Activities of Daily Living).The FAAM-ADL consists of 21 questions, with a maximum score of 4 per question. The sum of the scores of answered questions is divided by the highest potential score (84 if all 21 questions are answered) and converted to a total score out of 100, with a minimum score of 0. Higher scores indicate better function. Total score range is 0 to 100.
  units on a scale | 33.7 (14.1) | 46.8 (24.2) | 40.3 (19.1)

OUTCOME MEASURES:

1. Primary Outcome: Patient Reported Pain (VAS)
Description: Visual Analog Scale (0 - 100) to assess pain at various musculoskeletal sites. Patients are presented with a slider on a scale to indicate the degree to which they are experiencing pain on a scale from "No Pain" at the far left to "Worst Pain" at the far right. The position on the scale is then translated into a number from 0 (no pain) to 100 (worst pain).
Time Frame: 0-24 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Group I: Patients in Group I were assigned to receive a course of CAM walker boot treatment for a period of six weeks.
- Group II: Patients in Group II were assigned to receive a course of CAM walker boot treatment with an EVENup orthotic shoe lift to be worn on the contralateral foot for a period of six weeks.
Arm/Group | Group I | Group II
Number analyzed (Participants) | 3 | 3
score on a scale
  0 weeks - Lower Back | 0 (0) | 0 (0)
  0 weeks - Right Hip | 0 (0) | 0 (0)
  0 weeks - Left Hip | 11 (19.1) | 0 (0)
  0 weeks - Right Knee | 2 (3.5) | 0 (0)
  0 weeks - Left Knee | 0 (0) | 0 (0)
  0 weeks - Right Ankle | 12.7 (21.9) | 29.7 (30.5)
  0 weeks - Left Ankle | 15.7 (27.1) | 0 (0)
  0 weeks - Right Foot | 0 (0) | 26.7 (46.2)
  0 weeks - Left Foot | 3.7 (6.3) | 0 (0)
  6 weeks - Lower Back | 0 (0) | 0 (0)
  6 weeks - Right Hip | 0 (0) | 0 (0)
  6 weeks - Left Hip | 1.7 (2.9) | 3.3 (5.8)
  6 weeks - Right Knee | 2 (3.5) | 0 (0)
  6 weeks - Left Knee | 0 (0) | 16.7 (28.9)
  6 weeks - Right Ankle | 0 (0) | 3.3 (5.8)
  6 weeks - Left Ankle | 10.3 (17.9) | 0 (0)
  6 weeks - Right Foot | 0 (0) | 4.7 (8.1)
  6 weeks - Left Foot | 4 (6.9) | 0 (0)
  12 weeks - Lower Back | 0 (0) | 0 (0)
  12 weeks - Right Hip | 0 (0) | 0 (0)
  12 weeks - Left Hip | 0 (0) | 0 (0)
  12 weeks - Right Knee | 0 (0) | 0 (0)
  12 weeks - Left Knee | 0 (0) | 0 (0)
  12 weeks - Right Ankle | 7.7 (13.3) | 4.7 (8.1)
  12 weeks - Left Ankle | 6.7 (11.5) | 0 (0)
  12 weeks - Right Foot | 0 (0) | 5.7 (9.8)
  12 weeks - Left Foot | 2 (3.5) | 0 (0)
  24 weeks - Lower Back | 0 (0) | 0 (0)
  24 weeks - Right Hip | 0 (0) | 0 (0)
  24 weeks - Left Hip | 0 (0) | 0 (0)
  24 weeks - Right Knee | 0 (0) | 0 (0)
  24 weeks - Left Knee | 9.7 (16.7) | 0 (0)
  24 weeks - Right Ankle | 1.3 (2.3) | 0 (0)
  24 weeks - Left Ankle | 4 (6.9) | 0 (0)
  24 weeks - Right Foot | 0 (0) | 3.7 (6.4)
  24 weeks - Left Foot | 0 (0) | 0 (0)

2. Primary Outcome: Patient Reported Outcome (FAAM-ADL, 0 - 100)
Description: FAAM-ADL (Foot and Ankle Ability Measure - Activities of Daily Living, [0 -100]).The FAAM-ADL consists of 21 questions, with a maximum score of 4 per question. The sum of the scores of answered questions is divided by the highest potential score (84 if all 21 questions are answered) and converted to a total score out of 100, with a minimum score of 0. Higher scores indicate better function. Total score range is 0 to 100.
Time Frame: 0-24 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group I | Group II
Number analyzed (Participants) | 3 | 3
score on a scale
  0 weeks | 33.7 (14.1) | 46.8 (24.2)
  6 weeks | 59.9 (4.8) | 88.9 (8.1)
  12 weeks | 86.1 (14.8) | 97.2 (2.5)
  24 weeks | 92.9 (6.2) | 99.6 (0.7)

ADVERSE EVENTS:
Time Frame: Patients were monitored for the duration of their participation (24 weeks).
Description: The MGB Adverse Event Tracking Log was utilized.
Arm/Group | Group I: CAM Walker Boot | Group II: CAM+EVENup Orthotic Shoe Lift
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-17): https://cdn.clinicaltrials.gov/large-docs/63/NCT04164563/Prot_SAP_000.pdf